CLINICAL TRIAL: NCT04352452
Title: SOS - Save Our Surgeons - Differences in Musculoskeletal and Cognitive Stress of Robot-assisted Laparoscopic Surgery vs. Conventional Laparoscopic Surgery
Brief Title: Save Our Surgeons - Differences in Stress of Robot-assisted Laparoscopic Surgery vs. Conventional Laparoscopic Surgery
Acronym: SOSII
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Institute of Occupational and Social Medicine and Health Services Research, Tuebingen (Unknown)
Responsible Party: Sponsor
Other Study IDs: MT_SOS II
Record Dates: First submitted 2019-02-28; First posted 2020-04-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2022-11

CONDITIONS: Excessive Musculoskeletal Stress
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RALS: Surgeons perform robot-assisted laparoscopic surgery
  Interventions: Procedure: laparoscopic surgery
- CLS: Surgeons perform conventional laparoscopic surgery
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: laparoscopic surgery — differences in musculoskeletal and cognitive stress

SUMMARY:
Monocentric trial to evaluate differences in musculoskeletal and cognitive stress of robot-assisted laparoscopic surgery (RALS) vs. conventional laparoscopic surgery (CLS). Demographic and personal data are collected and pseudonymized as well as video recordings are performed during surgery. Simultaneously, surface electromyography (EMG) and electrocardiography (ECG), motion tracking data are collected. Additionally, saliva cortisol, perceived discomfort and mental load will be assessed within certain time intervals. The surgeon is not disturbed in his activity and movement by the equipment.

Afterwards, the surgeon will be interviewed in a 15-minute standardized interview about the surgery process and the subjective stress sensitivity. Only routine interventions will be recorded, in case of unforeseen complications, the recording will be stopped immediately

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 68 years
* Able to work in full shift
* trained surgeons in RALS and CLS
* written informed consent

Exclusion Criteria:

* persons influenced by analgesics or muscle relaxants
* not being able to work for any reason
* persons with acute diseases or pain Depending on the degree of severity, persons with diseases of the spine, hand-arm system, muscle disorders, symptomatic neurological-psychiatric disorders, when indicated regular medications, acute pain symptoms, diseases or other current illnesses must be excluded

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female gynecological surgeons who are experienced and must have performed a theoretical and virtual reality based training program in robotic assisted surgery.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Median muscular load of the bilateral trapezius pars descendens muscle surface electromyography. | 75 Minutes
  Muscle activity will be recorded using bipolar surface electromyography and is defined as the root-mean-square (RMS) of electrical muscle activity. Muscle activity will be normalized to an isometric voluntary maximum electrical activation (MVE) and the 50th percentile the normalized RMS will be calculated [percent MVE]
Static muscular load of the bilateral trapezius pars descendens muscle | 75 Minutes
  Muscle activity will be recorded using bipolar surface electromyography and is defined as the root-mean-square (RMS) of electrical muscle activity. Muscle activity will be normalized to an isometric voluntary maximum electrical activation (MVE) and the 10th percentile of the normalized RMS [percent MVE] will be calculated.
sustained muscular activity of the bilateral trapezius pars descendens muscle | 75 Minutes
  Muscle activity will be recorded using bipolar surface electromyography and is defined as the root-mean-square (RMS) of electrical muscle activity. Muscle activity will be normalized to an isometric voluntary maximum electrical activation (MVE) and the number of episodes (≥ 8min) of the normalized RMS above 0.5percent MVE [n] will be calculated.
Muscular rest time of the bilateral trapezius pars descendens muscle | 75 Minutes
  Muscle activity will be recorded using bipolar surface electromyography and is defined as the root-mean-square (RMS) of electrical muscle activity. Muscle activity will be normalized to an isometric voluntary maximum electrical activation (MVE) and the frequency [n] and relative duration [percent] of the normalized RMS lower than 0.5percent MVE will be calculated.

SECONDARY OUTCOMES:
Median muscular load of the bilateral extensor digitorum and flexor carpi radials muscles | 75 Minutes
  Muscle activity will be recorded using bipolar surface electromyography and is defined as the root-mean-square (RMS) of electrical muscle activity. Muscle activity will be normalized to an isometric voluntary maximum electrical activation (MVE) and the 50th percentile the normalized RMS will be calculated [percent MVE]
Static muscular load of the bilateral extensor digitorum and flexor carpi radials muscles | 75 Minutes
  Muscle activity will be recorded using bipolar surface electromyography and is defined as the root-mean-square (RMS) of electrical muscle activity. Muscle activity will be normalized to an isometric voluntary maximum electrical activation (MVE) and the 10th percentile of the normalized RMS [percentMVE] will be calculated.
sustained muscular activity of the bilateral extensor digitorum and flexor carpi radials muscles | 75 Minutes
  Muscle activity will be recorded using bipolar surface electromyography and is defined as the root-mean-square (RMS) of electrical muscle activity. Muscle activity will be normalized to an isometric voluntary maximum electrical activation (MVE) and the number of episodes (≥ 8min) of the normalized RMS above 0.5percent MVE [n] will be calculated.
Muscular rest time of the bilateral extensor digitorum and flexor carpi radials muscles | 75 Minutes
  Muscle activity will be recorded using bipolar surface electromyography and is defined as the root-mean-square (RMS) of electrical muscle activity. Muscle activity will be normalized to an isometric voluntary maximum electrical activation (MVE) and the frequency [n] and relative duration [percent] of the normalized RMS lower than 0.5percent MVE will be calculated.
Shoulder abduction angle [degree] | 75 Minutes
  Shoulder abduction angle will be assessed by the difference of two gravimetric position sensors placed on the upper back and the lateral side of the upper arm.
trunk flexion angle [degree] | 75 Minutes
  Trunk flexion angle will be assessed by the difference of two gravimetric position sensors placed on the upper and lower back.
head flexion angle [degreee] | 75 Minutes
  Head flexion angle will be assessed by the difference of two gravimetric position sensors placed on the upper back and the forehead.
Frequency of perceived physical discomfort [n] | 75 Minutes
  Subjects will be asked in 20-min intervals throughout the surgery whether they feel any discomfort [yes or no]
Intensity of perceived physical discomfort [0-10; 0 = nothing at all, 10 = extremely high | 75 Minutes
  Subjects will be asked in 20 -min intervals throughout the surgery about their level of perceived physical discomfort using a numeric rating scale [0 to 10].
Subjective mental demand [0 - 21; 0 = very low, 21 = very high] | 75 Minutes
  Subjective mental demands will be assessed by the mental demand subscale of the NASA TLX questionnaire
heart rate [beats per minute] | 75 Minutes
  Heart rate will be recorded by a one channel electrocardiogram
Heart rate variability as the Standard Deviation of NN intervals [ms] | 75 Minutes
  Heart rate will be recorded by a one channel electrocardiogram and the standard Deviation of the NN interval will be calculated
Heart rate variability as the Root Mean Squers of Successive Differences [ms] | 75 Minutes
  Heart rate will be recorded by a one channel electrocardiogram and the root mean square of the successive differences will be calculated

OTHER OUTCOMES:
Body height [cm] | 5 Minutes
  The Nordic Questionnaire will be used to determine subjects body height Physical activity [hours of sports per week work experience [years] musculoskeletal complaints in the last 12 month, last week, and point prevalence [n]
Body weight [kg] | 5 Minutes
  The Nordic Questionnaire will be used to determine subjects body weight
Physical activity [hours of sports per week] | 5 Minutes
  The Nordic Questionnaire will be used to determine subjects weekly physical activity
work experience [years] | 5 Minutes
  The Nordic Questionnaire will be used to determine subjects work experience
Musculoskeletal complaints in the last 12 month, last week, and point prevalence [n] | 5 Minutes
  The Nordic Questionnaire will be used to determine subjects musculoskeletal complaints in the last 12 month, last week, and point prevalence

CONTACTS AND LOCATIONS:
Overall Officials: Sara Brucker, Prof. Dr., Study Chair — Department of Women's Health, University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Department of Women's Health, Tübingen, Germany